CLINICAL TRIAL: NCT05674903
Title: Deep Brain Therapy With Low-intensity Ultrasound for Generalized Chronic Pain: A Pilot Study of Target Engagement and Analgesic Effects
Brief Title: Deep Brain Therapy With Low-intensity Ultrasound for Generalized Chronic Pain
Acronym: DBT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jan Kubanek, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00162656
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Widespread Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active stimulation (Experimental): Low-intensity transcranial focused ultrasound stimulation of deep brain targets involved in pain perception Intervention: Device: Diadem prototype
  Interventions: Device: Verum stimulation with Diadem prototype
- Sham stimulation (Sham Comparator): Low-intensity transcranial focused ultrasound stimulation using unfocused wave Intervention: Device: Diadem prototype
  Interventions: Device: Sham stimulation with Diadem prototype

INTERVENTIONS:
Device: Verum stimulation with Diadem prototype — Diadem prototype device delivers focused low-intensity ultrasound stimulation
  Arms: Active stimulation
Device: Sham stimulation with Diadem prototype — Diadem prototype device delivers active sham, unfocused low-intensity ultrasound stimulation
  Arms: Sham stimulation

SUMMARY:
This study will evaluate a new form of non-invasive deep brain therapy for individuals with generalized chronic pain. Low-intensity transcranial focused ultrasound stimulation will first be delivered using a range of stimulation parameters during psychophysical and physiological monitoring. A well-tolerated stimulation protocol will be selected for subsequent testing in a blinded randomized sham-controlled cross-over trial. The trial will evaluate brain target engagement using magnetic resonance imaging and CVAS and PROMIS numerical rating scales of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, any gender
2. Primary diagnosis of generalized chronic pain or widespread chronic pain.
3. Moderate-to-severe chronic pain lasting at least 2 months
4. Stated willingness to comply with all study procedures and avoid changes to current treatments (medications, physical therapy, cognitive behavioral therapy) for the duration of the study
5. For females of reproductive potential: negative pregnancy test or use of highly effective contraception for at least 1 month prior to baseline; agreement to use such a method throughout the study
6. Capacity to provide informed consent; provision of a signed and dated consent form

Exclusion Criteria:

1. History of serious brain injury or other neurologic disorder
2. Poorly managed general medical condition
3. Pregnant or breast feeding
4. Implanted device in the head or neck
5. MRI intolerance or contraindication
6. Brain stimulation (e.g., VNS, TMS) in the past month
7. Lifetime history of a serious suicide attempt (Hooley et al., 2014)
8. Clinically inappropriate for participation in the study as determined by the study team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Target engagement: brain activation | 1 day At MRI study visit
  MRI quantification of blood oxygenation level dependent (BOLD) activation.
Target engagement: brain connectivity | 1 day At MRI study visit
  Pearson's correlation of BOLD signals between the stimulated target and connected regions.
Pain intensity: momentary change | 1 day At stimulation visit
  Computerized Visual Analogue Scale. The scale is measured using a continuous slider. At its left boundary, the slider indicates no pain (score 0). At its right boundary, the slider indicates worst pain imaginable (score 100). A lower score indicates a better treatment outcome.
Pain intensity: subjective state | 1 day At stimulation visit
  PROMIS scale of pain intensity. Scores range from 1 (no pain) to 5 (severe pain). A lower score indicates a better treatment outcome.
Depression scale: subjective state | 1 day At stimulation visit
  PROMIS scale of depression. Scores range from 1 (not at all depressed) to 5 (severely depressed). A lower score indicates a better treatment outcome.
Anxiety scale: subjective state | 1 day At stimulation visit
  PROMIS scale of anxiety. Scores range from 1 (not at all anxious) to 5 (severely anxious). A lower score indicates a better treatment outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riis TS, Feldman DA, Losser AJ, Okifuji A, Kubanek J. Noninvasive targeted modulation of pain circuits with focused ultrasonic waves. Pain. 2024 Dec 1;165(12):2829-2839. doi: 10.1097/j.pain.0000000000003322. Epub 2024 Jul 30. PMID 39073370